CLINICAL TRIAL: NCT02382042
Title: Intensive Referral Intervention to Improve Substance Use Disorder Treatment Outcomes Among Rural and Highly Rural Veterans
Acronym: IRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen M. Grant, Principal Investigator, VA Nebraska Western Iowa Health Care System
Model: Parallel | Purpose: Treatment
Other Study IDs: N32-FY13Q1-S1-P00642
Record Dates: First submitted 2015-02-23; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Substance Use Disorders
Keywords: Rural Health; Veterans; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Referral Intervention (Active Comparator)
  Interventions: Behavioral: Intensive Referral Intervention
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Intensive Referral Intervention
  Arms: Intensive Referral Intervention

SUMMARY:
Background Participation in continuing care is one of the two most significant factors in preventing relapse after intensive Substance Use Disorder (SUD) treatment.1 A primary component of continuing care, social support, is a protective factor for SUD treatment relapse.2 Social support provided by community self-help groups (e.g. 12-step programs such as Alcoholics Anonymous) improves Substance Use Disorder (SUD) treatment outcomes.1,4 Post-treatment referral to self-help groups was recently described as "an effective, low-cost option,"3 but counselors vary in their referral methods, often simply telling patients to find and attend meetings in their community.

In a study of urban veterans leaving treatment, researchers increased 1-year SUD abstinence rates by more than 24% through a three-step intensive referral intervention.5 First, counselors discussed the importance of social support and meeting attendance. Second, counselors identified accessible self-help meetings near the SUD treatment site and arranged for a meeting liaison to accompany the patient to a meeting. Third, counselors followed up on attendance and addressed obstacles. A follow-up study found patients with co-morbid SUD and psychiatric problems significantly benefitted from the intervention.6

The investigators have adapted this intervention so that it can be utilized in a rural as well as urban setting. The investigators have trained clinical staff, measured their fidelity to the intervention and successfully implemented it across three Veteran's Affairs (VA) Substance Use Disorder (SUD) treatment programs (Omaha, Lincoln and Grand Island). In 2012 an intriguing study showed that peer referral to 12-step support groups was significantly more effective than clinician referral.7 This is of particular interest given the scarcity of addiction counselors in rural communities and enhances the intervention's applicability to rural settings and other disciplines.

Specific Aim The investigators propose implementing this intervention in a correction population (Intervention Group) and comparing outcomes between the Intervention Group and a group who are receiving standard correction services (Standard Group).

Methods Phase I: Adapt Intensive Referral Intervention for correction population Phase II: Train correction staff in Intervention Research staff will train and continue to monitor trained correction staff to ensure fidelity to intervention and provide feedback to staff and leadership regularly.

Phase III: Comparison between Intervention Group and Standard Group The two groups will be compared on measures of interest to the Nebraska Department of Correctional Services and on measures of substance use, support group attendance and involvement at standard time points.

DETAILED DESCRIPTION:
Rural veterans have disproportionately served in OEF and OIF and are returning to their communities with significant substance use disorder (SUD) and trauma-related symptoms. Participation in post-treatment continuing care is one of the two most significant factors in preventing relapse after intensive SUD treatment,1 but as a result of the reorganization of SUD services within the VHA, rural veterans have less access than non-rural veterans to continuing care. A primary component of continuing care, social support, is a protective factor for SUD treatment relapse2 and post-deployment traumatic stress symptoms.3 Social support provided by community self-help groups (e.g. 12-step programs such as Alcoholics Anonymous) improves outcomes1,4 and efforts to promote participation reduce continuing care costs.2 Post-treatment referral to self-help groups was recently described as "an effective, low-cost option,"3 but treatment counselors vary in their referral methods, often simply telling patients to find and attend meetings in their community.

In a study of urban veterans leaving treatment, researchers increased 1-year SUD abstinence rates by more than 24% through a three-step intensive referral intervention.5 First, counselors discussed the importance of social support and meeting attendance. Second, counselors identified accessible self-help meetings near the SUD treatment site and arranged for a meeting liaison to accompany the patient to a meeting. Third, counselors followed up on attendance and addressed obstacles. A follow-up study found patients with comorbid SUD and psychiatric problems (like Post Traumatic Stress Disorder) significantly benefitted from the intervention.6

Implementing intensive referral with rural veterans is problematic because their initial SUD treatment typically occurs in an intensive residential setting in a location which is removed from the veteran's home and family. During this intensive residential SUD treatment, rural veterans attend self-help meetings near the residential treatment program with the goals of 1) identifying meetings they enjoy, 2) developing relationships with others who attend these meetings, and 3) obtaining a sponsor who will serve as a mentor to the newly sober veteran. However, upon discharge from residential SUD treatment, rural veterans return to their rural communities without these supports in place. Additionally, rural veterans attending 12- step meetings are likely to have challenges unique to their rural settings. In rural communities veterans are more likely to be recognized by others they know and rural residents rate self-help groups as less acceptable than urban residents do.7 Additionally, the only self-help groups consistently available in small communities are AA meetings which may cause some tension and ambivalence in those with problems other than alcohol.

Family members are another source of social support preventing SUD relapse,8 but rural veterans may not receive the same family support benefits urban veterans do. In urban veterans' SUD treatment, family members are typically involved in their treatment. The family members of rural veterans, however, are less likely to attend educational, individual or group sessions given their distance from the residential SUD treatment site and typically have no support themselves as they interact with their returning veteran. Thus, rural veterans return home to live with families who may be less able to provide meaningful support to their newly sober veteran.

Further complicating this clinical picture is the presence of trauma symptoms. Among those seeking SUD treatment, nearly all report lifetime trauma exposure and one-third are diagnosed with post-traumatic stress disorder (PTSD).9 The prevalence among veterans is likely higher. Persons with dual disorders, such as PTSD and SUD, have poorer SUD treatment outcomes, and may be at higher risk for homelessness. Self-help groups improve the outcomes for those with concurrent PTSD and SUD.10 Dr. Timko's work has established that the intensive referral intervention, to be adapted in this project, resulted in an 18% reduction in the number of psychiatric symptoms and a 26% reduction in perceived need for mental health treatment.6

The investigators propose an intensive referral adapted to the needs of rural veterans, modifying the existing intensive referral two ways. First, the adapted intensive referral will present information addressing recovery challenges specific to rural veterans: building support networks, overcoming distance, finding transportation, locating professional resources, using online support, and preparing for relapse emergencies. These modifications will also be provided as options for those accessing the VA's intensive referral Self-Help Toolkit, available online. Second, the adapted intensive referral will enlist family support for self-help groups, stressing the importance of meetings and encouraging family members to provide transportation and/or attend the meetings.

Purpose and Objectives:

The purpose of this project is to adapt an intensive self-help referral intervention for the 450 rural and highly rural veterans in SUD treatment in NWI HCS, train one-half of the Nebraska Wwesterion Iowa Health Care System SUD treatment staff in the intervention and test it as a pilot project. The Specific Aims of the project are:

1. To determine whether adapted intensive referral to community-based support groups increases the effectiveness of SUD treatment in rural veterans,
2. To determine if co-occurring PTSD and family involvement are factors in responsiveness to the adapted intensive referral intervention.

Methodology:

Phase I: Intensive Referral Self-Help Toolkit Adapted to Serve Rural Veterans The investigators will adapt the VA's Intensive Referral Self-Help Toolkit, a practical guide to assist veterans' transition into community self-help groups. The adaptation will specifically address factors which are unique to rural veterans such as lack of "drug-related" meetings, concerns about anonymity, distance and transportation. Secondly, the intensive referral will be adapted to include the enhancement of family involvement in the referral process. Dr. Timko will assist us with the adaptation and feedback from veterans, family members, 12-step group liaisons and providers will inform modification of the Toolkit to address the specific needs of rural veterans, their families, and their healthcare providers. Also in Phase I the Project Peer Support Specialist will canvass self-help groups throughout rural Nebraska and western Iowa to identify 12-step meetings which are welcoming to persons with drug as well as alcohol addictions and individuals willing to serve as a group liaison to support and attend meetings with the veteran and their family member.

Phase II: SUD Staff Trained in Intervention Dr. Grant and the Project Manager will meet with SUD treatment leadership and staff at the three Nebraska-Western Iowa Health Care System (NWI-HCS) locations (Grand Island, Lincoln and Omaha) and orient them to the project. One-half of the Addiction Therapists at each site will be trained in the modified Intensive Referral Self-Help Toolkit in Year One. These Addiction Therapists will role-play this intervention with Project staff in individual and group settings. The remaining Addiction Therapists will continue to utilize Standard Referral (i.e. simply encouraging meeting attendance). The Program Manager will continue to monitor those trained Addiction Therapists to ensure that the intervention remains consistent with the Toolkit and will meet with staff and leadership regularly at each site to provide feedback. Veterans assigned to trained Addiction Therapists will receive Intensive Referral while those assigned to other Addiction Therapists will receive Standard Referral.

Phase III: Comparison Between Intensive Referral Group and Standard Care Group Rural veterans will be contacted by telephone at 6-months post discharge from intensive SUD treatment. The two groups (Intensive Referral v. Standard Referral) will be compared on measures of substance use, addiction severity, trauma symptoms, satisfaction with referral process, family support, support group attendance and involvement.

Summary of data analysis and statistical methods:

Study participants will be contacted by telephone at 6-months post discharge from intensive SUD treatment. The two groups (Intensive Referral v. Standard Referral) will be compared on measures of substance use, addiction severity, trauma symptoms, family support, support group attendance and involvement and satisfaction with the referral process. The investigators also will determine whether veterans with a co-occurring PTSD diagnosis benefit more from the enhanced intensive referral compared to standard referral and the investigators will determine whether 6-month abstinence rates are lower for those with family support compared to those without family support.

While the populations of interest for this study are rural and highly rural Veterans, rural and highly rural status will be defined by zip code of residence at the time the follow-up questionnaire is administered, six months after discharge from SUD treatment. Patients may be admitted from a 'rural zip code' but at discharge move to a residence in an 'urban zip code.' The investigators will initially compare outcomes between all participants who received the Intensive Referral and those who received Standard Referral. The investigators will then compare outcomes between the two groups (Intensive Referral v. Standard Referral) in those veterans who are living in rural or very rural zip codes at six months post-discharge.

In order to compare two groups of veterans (those who received Intensive Referral and those who received Standard Referral), a series of independent sample t-tests will be run to see whether these two groups significantly differ on measures of substance use, addiction severity, trauma symptoms, satisfaction with referral process, and family support. Next the investigators will use Pearson correlation coefficients to look for significant positive or negative effects of referral type (i.e., intensive v. standard) with the measures listed above. The next step of the process will be to run ordinary least squares (OLS) regression models given the continuous nature of our main outcome variable, substance use. The investigators will first run models to examine main effects. Next, the investigators will test for interaction effects to determine whether the effect of PTSD on substance use disorder varies by type of referral. Finally, ordinary least squares regression models will be run to determine whether 6-month abstinence rates are lower for those without family support compared to those with family support.

Innovation:

To our knowledge, this will be the first evidence-based substance abuse intervention to be modified for rural veterans. If effective, this SUD intervention will be the first to:

* Specifically improve sobriety rates in rural veterans,
* Incorporate family members into the intervention,
* Assess rural veteran satisfaction with the intensive referral,
* Determine if trauma symptoms are improved in rural veterans with adapted intensive referral,
* Determine if family involvement enhances responsiveness to adapted intensive referral, and
* Significantly decrease relapse rates in rural veterans, thus decreasing their re-hospitalizations and subsequent health care costs.

ELIGIBILITY:
Inclusion Criteria:

* All Veterans in SUD residential and outpatient treatment facilities in Grand Island, Lincoln and Omaha VA sites who are able to provide informed consent will be eligible for this research study.
* Eligibility to provide informed consent will be determined by completing the MINI-COG, a brief 3-minute instrument to screen for cognitive impairment.

Exclusion Criteria:

-If the patient is cognitively impaired, as determined by the MINI-COG, he/she will not be eligible for study participation.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Sobriety | 6 months
  Levels of sobriety will be measured by utilizing a time line fall back calendar.This measure outlines when the amount and timeline that a participant has used a particular substance.